CLINICAL TRIAL: NCT00276068
Title: Vulvar Vestibulitis Trial: Desipramine-Lidocaine
Brief Title: Vulvar Vestibulitis Clinical Trial: Desipramine-Lidocaine
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rochester (Other)
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: 5R01HD040123-03 (NIH); 5R01HD040123-03 (NIH)
Record Dates: First submitted 2006-01-11; First posted 2006-01-12 (Estimated); Last update posted 2007-11-14 (Estimated); Status verified 2007-11

CONDITIONS: Vulvar Disease
Keywords: Vulvar vestibulitis; Vulvodynia; Desipramine; Lidocaine; Genetics
MeSH Terms: conditions — Vulvar Diseases; Vulvar Vestibulitis; Vulvodynia | interventions — Lidocaine; Desipramine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: topical lidocaine + oral desipramine, and/or placebo

SUMMARY:
The Vulvar Vestibulitis Clinical Trial (VVCT) a randomized, placebo-controlled, double blinded clinical trial. We will study the clinical efficacy of four medical treatments for vulvar vestibulitis: topical lidocaine, oral desipramine, combined lidocaine and desipramine, and placebo cream and capsules. Desipramine is a tricyclic antidepressant commonly used by clinicians for treatment of several chronic pain conditions that demonstrates an optimal side effect profile compared to other tricyclic antidepressants. Topical lidocaine has also been found to be beneficial for vulvar vestibulitis treatment in small studies. It is hypothesized that the combined use of oral desipramine and topical lidocaine will be more therapeutically effective than either one by itself and better than placebo.

DETAILED DESCRIPTION:
The Vulvar Vestibulitis Clinical Trial (VVCT) is a randomized, placebo-controlled, double-blinded clinical trial to study the clinical efficacy of four medical treatments for vulvar vestibulitis: 1) topical lidocaine, 2) oral desipramine, 3) combined lidocaine and desipramine, and 4) placebo cream and capsules. The duration of study drug will last 12 weeks with post-intervention follow-up at 6 and 12 months. We plan to enroll 128 subjects from the university-based clinical program at the University of Rochester (UR).Primary outcome variable will compare the reported pain of the "Tampon Test" (mean of Weeks -2, -1, and 0), prior to randomization to the reported pain of "Tampon Test" (mean of Weeks 10, 11, and 12). The dependent (primary outcome) variable will be defined as the percent change of mean "Tampon test" pain of Weeks (10, 11, and 12) from Weeks (-2, -1 and 0). The primary analysis of this 2X2 factorial design will involve fitting an Analysis of Covariance (ANCOVA) regression model to the percent change of mean "Tampon test" pain with the two treatment variables as the predictors while adjusting for the covariate age. We will test if the interaction between the two treatments in the ANCOVA model is significant at the .05 level. If the interaction effect is not significant, it will be dropped from the model and the conclusion will be drawn from the model with main effects only. If significant, the model with interactions will be adopted. SAS PROC GLM will be used in the analysis.

In the case of non-significant interaction, the primary analysis will be based on the ANCOVA model with main effects of treatments and adjusting for age. Since there are two treatments under investigation, the primary analysis will use the Bonferroni correction, i.e. will set alpha level of 0.025 (two-sided) to determine statistical significance. The significance of the main effect of each treatment will be assessed by t-tests in the ANCOVA model. The aim of the primary analysis is to determine whether each treatment is superior to placebo, and if both hypotheses hold, the double treatment therapy will be most effective under the additive effect assumption of the ANCOVA model. The ANCOVA model compares all subjects who receive that treatment with all subjects who do not, irrespective of whether they receive the other treatment, after adjusting for the other treatment and age of subject, and is more powerful in finding individual treatment effects in the study.

If interaction between treatments is significant, the ANCOVA model with interaction will estimate the treatment effects for each of the four groups. This model is able to test all 6 contrasts between the four combinations. A hierarchical (gatekeeping) testing strategy to maintain a family-wise error rate will be adopted as the following: the first stage will compare desipramine or lidocaine individually to placebo with multiplicity-adjusted p-values. If a significant difference (one or both null hypotheses rejected) is found for either or both individual agents, then the analysis will proceed to the second-stage of hypothesis which will compare the effects of the active desipramine/active lidocaine treatment to the double placebo. If a significant difference (null hypothesis rejected) is found for combined therapy over placebo based on the multiplicity-adjusted p-value, then the final (tertiary) stage of comparison will be performed comparing combined therapy to individual therapy. In the hierarchical (gatekeeping) testing procedures, inferences in each stage depend on the acceptance or rejection of null hypotheses in all previously stages, and each stage serves as a gatekeeper for the stages later in the sequence. In our strategy for the model with significant interaction effect, if at least one hypothesis has been rejected, then the next stage of hypotheses will be tested, and the family-wise error rate is controlled at the .05 level.

Secondary analyses will include subset analysis, comparison of the double-active treatment group against the others (placebo and the single-treatment groups) on percent change of mean "Tampon test" as well as standardized pain measures such as the Brief Pain Inventory and the McGill Pain Questionnaire. This is to explore if the active desipramine/active lidocaine treatment has more advantages that may not be shown in the ANCOVA model. The secondary analysis is to explore supportive evidence to the primary objective of this trial, and no confirmatory conclusions are needed. In the secondary analysis, confidence intervals and statistical tests are of exploratory nature and no claims are intended.

Primary and secondary outcome variables will be analyzed according to a modified "intention to treat" with "last observation carried forward". The sample analyzed for the primary outcome will include the first three or fewer pre-randomization Tampon Test measures and the last three or fewer post-randomization Tampon Test measures, up to and including study Week 12. The subject sample analyzed for drug safety/side effects will include all subjects who have taken at least one dose of study drug.

ELIGIBILITY:
Inclusion Criteria: Candidates must report greater than three continuous months' duration of vulvar symptoms of insertional dyspareunia, pain with tampon insertion, or pain to touch.

Physical exam should demonstrate "Friedrich's Criteria" which includes Criterion #1: history of severe pain on vestibular touch or attempted vaginal entry for a continuous duration of 6 months or greater. Criterion #2: tenderness localized within the vestibule.

The candidate should not demonstrate any other specific neuropathology Pre-randomization laboratory testing should fail to identify atrophic vaginitis, dermatitis such as vulvar dystrophy, or pathogens such as fungus, or herpes.

The candidate should not report use tricyclic-class or topical lidocaine within 30 days of the study.

Candidates will need to be capable of keeping adequate records and demonstrate reliability in use of medication.

If the candidate is premenopausal, adequate contraception will be necessary including oral contraceptives, barrier method, progestational contraceptives, vasectomy, tubal ligation, and hysterectomy.

Exclusion Criteria:

History of cardiac arrhythmia, syncopal episodes, seizures, vulvar cancer, specific dermatoses, choreoathetosis or major depression.

Active infection with herpes simplex, herpes zoster, Bartholin's abscess, Pregnancy, Active liver disease or renal disease, Evidence on prior vulvar biopsy or clinical impression of specific vulvar dermatoses such as lichen sclerosus, squamous cell hyperplasia, or lichen planus Positive culture for fungus (persistence of pain after treatment of particular infection and negative culture will not exclude subject from the study) Known hypersensitivity to either active agents (desipramine/lidocaine) or cream vehicle (Moisturelle cream) Immunocompromised state, History of illicit drug or alcohol abuse within the last year Serious or unstable medical or psychiatric conditions, Evidence of conduction abnormalities (especially prolonged QT interval) on ECG.

-

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 128 (Estimated)
Dates: Start 2002-08; Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
Primary outcome variable will compare the reported pain of the "Tampon Test" (mean of Weeks -2, -1, and 0), prior to randomization to the reported pain of "Tampon Test" (mean of Weeks 10, 11, and 12). | The dependent (primary outcome) variable will be defined as the percent change of mean "Tampon test" pain of Weeks (10, 11, and 12) from Weeks (-2, -1 and 0).

SECONDARY OUTCOMES:
24 hour mean pain score | Weeks (10, 11, and 12) from Weeks (-2, -1 and 0)
frequency of intercourse | Weeks (10, 11, and 12) from Weeks (-2, -1 and 0)
intensity of intercourse pain | Weeks (10, 11, and 12) from Weeks (-2, -1 and 0)
selected psychometric tests
quantitative pain level measured by the Vulvar Algesiometer / Cotton Swab Test
side-effects | The subject sample analyzed for drug safety/side effects will include all subjects who have taken at least one dose of study drug.
Interleukin 1 RA and MC1-R polymorphisms

CONTACTS AND LOCATIONS:
Overall Officials: David C Foster, MD, MPH, Principal Investigator — University of Rochester
Locations (1):
- Strong Memorial Hospital, Rochester, New York, United States

REFERENCES:
- [Derived] Foster DC, Kotok MB, Huang LS, Watts A, Oakes D, Howard FM, Poleshuck EL, Stodgell CJ, Dworkin RH. Oral desipramine and topical lidocaine for vulvodynia: a randomized controlled trial. Obstet Gynecol. 2010 Sep;116(3):583-593. doi: 10.1097/AOG.0b013e3181e9e0ab. PMID 20733439
- [Derived] Foster DC, Beth Kotok M, Huang LS, Watts A, Oakes D, Howard FM, Stodgell CJ, Dworkin RH. The tampon test for vulvodynia treatment outcomes research: reliability, construct validity, and responsiveness. Obstet Gynecol. 2009 Apr;113(4):825-832. doi: 10.1097/AOG.0b013e31819bda7c. PMID 19305326